CLINICAL TRIAL: NCT05549024
Title: 68Ga-RM26-RGD PET/CT Imaging in the GRPR and αvβ3 Positive Tumor Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-RR
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Prostate Cancer; Brain Tumor; PET/CT Imaging
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Brain Neoplasms | interventions — Fluorodeoxyglucose F18; 68Ga-NOTA-RM26

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 68Ga-RM26-RGD and 18F-FDG PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-RM26-RGD and 18F-FDG, respectively.
  Interventions: Drug: 68Ga-RM26-RGD; Drug: 18F-FDG
- 68Ga-RM26-RGD and 68Ga-RM26 PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-RM26-RGD and 68Ga-RM26, respectively.
  Interventions: Drug: 68Ga-RM26-RGD; Drug: 68Ga-RM26
- 68Ga-RM26-RGD and 68Ga-RGD PET/ CT scan (Experimental): Within 2 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-RM26-RGD and 68Ga-RGD, respectively.
  Interventions: Drug: 68Ga-RM26-RGD; Drug: 68Ga-RGD

INTERVENTIONS:
Drug: 68Ga-RM26-RGD — Intravenous injection of 68Ga-RM26-RGD with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/ kg.
  Other Names: 68Ga-RM26-RGD injection
Drug: 18F-FDG — 18F-FDG injection
  Other Names: Intravenous injection of 18F-FDG with a dosage of approximately 3.7-5.55 MBq (0.1-0.15 mCi)/kg.
  Arms: 68Ga-RM26-RGD and 18F-FDG PET/ CT scan
Drug: 68Ga-RM26 — Intravenous injection of 68Ga-RM26-RGD with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/ kg.
  Other Names: 68Ga-RM26 injection
  Arms: 68Ga-RM26-RGD and 68Ga-RM26 PET/ CT scan
Drug: 68Ga-RGD — Intravenous injection of 68Ga-RGD with a dosage of approximately 1.8-2.2 MBq (0.05-0.06 mCi)/ kg.
  Other Names: 68Ga-RGD injection
  Arms: 68Ga-RM26-RGD and 68Ga-RGD PET/ CT scan

SUMMARY:
Based on the high expression of specific receptors on the surface of diseased tissues and neovascularization, noninvasive targeted molecular imaging can be used to visualize lesions in vitro by combining specific ligands labeled with short half-life isotopes. In this study, a novel dual-target imaging agent 68Ga-RM26-RGD was used for clinical study of tumor PET/CT imaging to further verify its clinical application value.

DETAILED DESCRIPTION:
Conventional 18F-FDG PET/CT has important diagnostic value in cell metabolism level, early metastasis, judging malignant potential and prognosis of tumors. It has been routinely used for staging and restaging of most tumors, but there are still some tumors with low uptake of 18F-FDG PET/CT. Receptor imaging with a single target also has some limitations in clinical application. For example, not all diseased cells express a large amount of single receptor on the surface, which greatly affects the judgment of the nature of the lesion. The dual-target molecular imaging based on GRPr expressed in the lesion site and integrin αvβ3 receptor highly expressed on the surface of the lesion neovascularization will overcome the above limitations and make full use of the advantages of the dual-target molecular imaging, which will greatly assist the diagnosis of malignant tumors such as breast\brain\prostate tumor which have high GRPr and αvβ3 receptor expression . In this study, a novel dual-target imaging agent 68Ga-RM26-RGD was used for PET/CT imaging of breast\brain\prostate cancer, compared with conventional 18F-FDG, or single target imaging agent 68Ga-RGD or 68Ga-RM26 PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed or suspected breast/brain/prostate cancer;
* 68Ga-RM26-RGD and 18F-FDG(or 68Ga-RM26 or 68Ga-RGD) PET/CT within 2 week;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance1 | through study completion, an average of 1 year
  comparing the SUV and number of primary or metastasis lesions detected by 68Ga-RM26-RGD and 18F-FDG PET/CT
Diagnostic performance2 | through study completion, an average of 1 year
  comparing the SUV and number of primary or metastasis lesions detected by 68Ga-RM26-RGD and 68Ga-RM26 PET/CT
Diagnostic performance3 | through study completion, an average of 1 year
  comparing the SUV and number of primary or metastasis lesions detected by 68Ga-RM26-RGD and 68Ga-RGD PET/CT

SECONDARY OUTCOMES:
The dosimetry of 68Ga-RM26-RGD | through study completion, an average of 1 year
  Measure the distribution of 68Ga-RM26-RGD in GRPR and αvβ3 positive tumor patients by 2-hour dynamic PET/CT acquisition by dosimetry software
68Ga-RM26-RGD uptake at different tumors | through study completion, an average of 1 year
  The SUV uptake of tumors and metastases in patients with breast/brain/prostate cancer was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China